CLINICAL TRIAL: NCT03574701
Title: Intranasal Retinoic Acid Treatment for Patients With Olfactory Loss: A Randomized Controlled Trial
Brief Title: Intranasal Retinoic Acid Treatment for Patients With OlfactoryLOSS: A RANDOMIZED CONTROLLED TRIAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Director, St. Paul's Sinus Centre, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H15-02095
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Olfactory Disorder
Keywords: olfactory; Vitamin A; Olfactory training; CRS
MeSH Terms: conditions — Anosmia | interventions — Vitamin A; Oils, Volatile

STUDY DESIGN:
Intervention Model Description: The patients will be randomized into 3 groups using the sealed envelope method. Each patient will be his or her own control. There will be two possible scenarios resulting from randomization:
  * Group A: This study group will receive intranasal vitamin A at 10,000 I.U. per day and olfactory retraining using scented oils in addition to their standard of care.
  * Group B: This study group will receive Vitamin A in addition to their standard of care. They will not receive olfactory retraining.
  * Group C: This study group will receive only standard of care .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A: Vitamin A and Olfactory Retraining (Experimental): Group A: This study group will receive intranasal vitamin A at 10,000 I.U. per day and olfactory retraining using scented oils in addition to their standard of care.
  Interventions: Dietary Supplement: Vitamin A
- B: Vitamin A (Experimental): Group B: This study group will receive Vitamin A in addition to their standard of care. They will not receive olfactory retraining.
  Interventions: Dietary Supplement: Vitamin A
- C: Standard of Care (No Intervention): Group C: This study group will receive only standard of care .

INTERVENTIONS:
Dietary Supplement: Vitamin A — The use of Vitamin A , in the treatment of olfactory loss has been previously studied in both animals and humans. These studies have shown promising results in the treatment of olfactory loss.
  Other Names: Essential oils
  Arms: A: Vitamin A and Olfactory Retraining; B: Vitamin A

SUMMARY:
About One to 2 percent of the North American population below the age of 65 years experience olfactory loss to a significant degree. It can result from advanced age, Post-infestious/inflammatory disorders, Obstructive disorders (e.g. nasal polyposis, tumors), posttraumatic (head trauma) and neurodegenerative disorders. Only a few studies have shown benefits of specific therapy for olfactory loss.

Vitamin has shown promise from both animal and human studies. However, none has studied the benefits of topical application of vitamin A. This study will be the first to examine this effect.

DETAILED DESCRIPTION:
1. Purpose

   To determine if there is an improvement in olfactory function following the use of intranasal Vitamin A in patients with post-inflammatory and/or post-traumatic olfactory loss.
2. Hypothesis

   There a significant improvement in olfactory function in patients with olfactory loss using intranasal vitamin A when compared with patients with olfactory loss not using intranasal vitamin A

   Null Hypothesis There is no significant improvement in olfactory function in patients with olfactory loss using intranasal vitamin A when compared with patients with olfactory loss not using intranasal vitamin A
3. Justification

   To treat post inflammatory and post-traumatic olfactory loss, a few controlled studies have shown a positive effect of a specific therapy for olfactory loss, such as olfactory training (using repeated intensive stimulation of the olfactory system and the use of prednisone. Other drugs studied like Vitamin B and Zinc, have either been insufficiently studied or showed no significant effect on olfactory loss.

   The use of Retinoic acid (Vitamin A), a fat-soluble vitamin, in the treatment of olfactory loss has been previously studied in both animal and human models and showed promise. However, no study has examined the use of topical administration of vitamin A. This study will be the first to examine this effect.
4. Objectives

   Primary Objective To determine if there is an improvement in olfactory function following the use of intranasal Vitamin A in patients with post-inflammatory and/or post-traumatic olfactory loss.

   Secondary Objectives To determine if patient quality of life is improved/affected by the use of intranasal vitamin A.
5. Research Method This is a Single blind Randomized Control Trial.

   Procedure

   The study population will be consecutive patients diagnosed with loss of olfactory function. It will be a single blind randomized control trial. Allocation concealment will be ensured by the use of sequentially numbered, opaque, sealed envelopes. An assessor blinded to which patient is using vitamin A will assess the primary outcome.

   Consent will be obtained for this study following diagnosis of the patient. After diagnosis, the patient will be sent a consent form and will be recruited on the next clinic visit.

   Screening: After diagnosis, there will be a screening period; inclusion/exclusion criteria for the study participation will be checked. Subjects who satisfy these criteria will be invited to participate in the study. The consent forms will be sent to them via email and their consent will be recorded.

   Blinding: The study will be single-blinded study. The patients will be randomized into 3 arms/groups. An assessor blinded to which patient is using vitamin A will assess the primary outcome.

   Study Arms/Groups: The patients will be randomized into 3 groups using the sealed envelope method. Each patient will be his or her own control. There will be two possible scenarios resulting from randomization:
   * Group A: This study group will receive intranasal vitamin A at 10,000 I.U. per day and olfactory retraining using scented oils. Olfactory retraining is a validated and effective method of improving olfaction in patients with olfactory loss and is currently being used at our centre as standard of care. It involves smelling 4 scented oils for 40 minutes everyday for the duration of the study. This is performed by the patients. They will also receive their standard of care budesonide (Pulmicort) for their sinonasal disease. The Vitamin A will be mixed with the budesonide and applied using the mucosal atomization device (MAD). This is a device used to apply intranasal medication. It reduces the medication to tiny droplets so they can reach all parts of the nose and sinuses.
   * Group B: This study group will receive Vitamin A and budesonide only. They will not receive olfactory retraining. These will also be applied using the MAD
   * Group C: This study group will receive only standard of care budesonide. The medication will also be applied using the MAD.

   Patients will also continue to receive all other standard of care medication and procedures as necessary.
6. Statistical Analysis

Sample size calculations According to the study conducted by Hummel et al, a the mean olfactory test (TDI) score was 19 with a standard deviation of 6.4. In order to have an 80% chance of detecting a clinically significant 6 point improvement in olfactory test (TDI) scores at a significant level of 5%, 108 patients will be required. This will be 36 patients per group. There is an approximately 10% drop out rate in studies conducted at the St Paul's sinus centre. Accounting for this drop out rate, a total of 120 participants (40 participants per group) will be required to conduct the study.

Statistical Comparisons Descriptive analysis will be used to describe demographic and some clinical outcomes. Mean, median and standard deviations will be used to describe these outcomes. The primary objective of this study is to compare olfactory function before and after the respective interventions among participants in the three groups. The dichotomous and continuous outcomes will be analyzed using Pearson Chi-squared test and analysis of variance (ANOVA). Analysis of variance will also be used to compare the olfactory test scores between the 3 groups and paired t-test for evaluating for statistical within the groups. Probability values less than 5% (α=0.05) will be considered significant. Sub-analysis by etiology of olfactory loss will also be done using the same methods.

ELIGIBILITY:
Inclusion Criteria:

Patients 19 years and above diagnosed with loss of olfactory function, (with or without history of sinonasal surgery) currently receiving sinonasal-related care at the St Paul's Sinus Centre.

Exclusion Criteria:

* Patients with Primary anosmia.
* Patients with baseline olfactory test scores >30 using Sniffin sticks test.
* Patients with sinonasal tumors
* Patients with polyps or significant inflammation blocking access of medication to the olfactory cleft.
* Patients allergic to topical Vitamin A
* Cystic fibrosis or syndromic patients
* Patients with autoimmune diseases that have sinus manifestations or affect sinus function
* Patients with previous history of hypervitaminosis A
* Patients with Neurological Disease (e.g. stroke history, Parkinson's disease)
* Patients who are pregnant

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-05-25 (Actual); Primary Completion 2021-12-25 (Estimated); Study Completion 2022-12-25 (Estimated)

PRIMARY OUTCOMES:
Olfactory Tests. | For each subject this test will take 30 minutes
  These tests will be performed by same blinded assessor using the "Sniffin sticks" kit described above. The test is divided into three subtests including tests for olfactory thresholds (using phenyl ethyl alcohol), odor discrimination, and odor identification (TDI). The sum of the three scores reliably indicates the degree of olfactory function.

SECONDARY OUTCOMES:
Sinonasal Outcomes Test - 22 (SNOT-22) | For each subject this test will take between 5-10 minutes.
  The SNOT-22 is a sinus-specific questionnaire that evaluates subjective symptoms for patients suffering from chronic rhinosinusitis. SNOT-22 is scored out of 110 (22 questions, up to 5-points each) has demonstrated internal consistency, reliability, discriminate and concurrent validity and responsiveness to change. Responses will be summated and considered as a continuous, numerical variable. Mean, median, standard deviation and inter-quartile range will be reported.
Sinus Mucosal Inflammation - Philpott-Javer (PJ) and Modified Lund-Kennedy (MLK) Endoscopic Staging System (ESS) | For each subject this test will take about 5 minutes.
  Sinonasal mucosal inflammation is an objective measure assessed endoscopically and graded on both the PJ and MLK ESS for CRS. This is a standard of care procedure at all clinic visits. Similar to the MLK ESS, the PJ ESS scores the sinus cavities as a collective based on endoscopic findings and the presence or absence of allergic mucin. Images and/or videos of all sinuses are captured at each visit and archived on the hospital network as a standard of care.
Questionnaire of Olfactory Disorders | For each subject this test will take about 10 minutes.
  The consists of 25 statements that were divided into three general domains: 17 negative statements (QOD-NS), two positive statements (QOD-PS), and six socially desired statements (QOD-SD). Negative statements give information about the degree patients suffer from olfactory impairment, whereas positive statements indicate how well patients cope with their olfactory deficit. Socially desired statements indicate the extent to which an individual's answers were credible, or whether the person was trying to create a certain impression by providing socially desirable responses. In addition there are also problem questions and questions regarding sense of smell on a visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Amin Javer, MD FRCSCFARS, Principal Investigator — University of British Columbia
Locations (2):
- Canada (2):
  - St Paul Hospital, Vancouver, British Columbia
  - St Paul Sinus Centre, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Undecided